CLINICAL TRIAL: NCT04361864
Title: Cross-sectional Survey on Patients With Urinary Tract Infections in Puy-de-Dôme : Epidemiology of Recurrent Urinary Tract Infections and Risk Factors
Acronym: IUR63
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Caisse Primaire d'Assurance Maladie du Puy-de-Dôme (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNI 2019 LESENS; 2019-A02703-54 (Other: 2019-A02703-54)
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RUTI: patients with at least 3 episodes of UTI during 2019
- UTI: patients with one or two episodes of UTI during 2019

SUMMARY:
Urinary tract infections (UTI) are an important part of infectious diseases. For some patients, those infections are recurrent and have many consequences such as altered quality of life, recurrent symptoms, antibiotics overuse… The primary purpose of this study is to estimate the proportion of patients in Puy-de-Dôme with recurrent urinary tract infections among patients with at least one UTI during 2019. The secondary purposes are : characteristics of patients with recurrent UTI, by sex ; determine predictive factors of recurrent UTI, by sex ; describe bacterial ecology of recurrent UTI and the proportion of multi-resistant bacteria.

ELIGIBILITY:
Inclusion Criteria:

* patient from 18 years old
* affiliated to the french healthcare system
* with at least one urinary tract infection during year 2019
* has accepted email contact with CPAM 63 (Caisse Primaire d'Assurance Maladie du Puy-de-Dôme)

Exclusion Criteria:

* pregnancy during year 2019
* none urinary tract infection reported in 2019

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with at least one urinary tract infection during year 2019
Sampling Method: Non-Probability Sample
Enrollment: 561 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Proportion of recurrent urinary tract infections | During year 2019
  Proportion, with its 95% confidence interval, of recurrent urinary tract infections, by sex, in the population of Puy-de-Dôme who reported having had at least one urinary tract infection in the year 2019.
  The diagnosis of recurrent urinary tract infection will be at least 3 urinary tract infections in one year

SECONDARY OUTCOMES:
age in year | day 1
  Risk factors of recurrent urinary tract infections
sexe | day 1
  Risk factors of recurrent urinary tract infections
, medical and surgical history | day 1
  Risk factors of recurrent urinary tract infections
life habits | day 1
  Risk factors of recurrent urinary tract infections
number of visits at the general practitioner | during year 2019
  measure of healthcare consumption with the number of visits at the general practitioner performed
number of urinalysis | during year 2019
  measure of healthcare consumption with the number of urinalysis performed
number of antibiotic therapies | during year 2019
  measure of healthcare consumption with the number of antibiotic therapies performed
quality of life | during year 2019
  quality of life evaluated with a self-reported questionnaire inspired by the Leicester Impact Scale
bacteriological characteristics of recurrent urinary tract infections | during year 2019
  evaluated with results of urinalysis, bacterial identification and antimicrobial susceptibility

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lesens, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France